CLINICAL TRIAL: NCT05249920
Title: Treatment of Acute Ischemic STroke With Edaravone Dexborneol Ⅱ (TASTE-2)
Brief Title: Treatment of Acute Ischemic STroke With Edaravone Dexborneol II (TASTE-2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yongjun Wang, President of Beijing Tiantan Hospital, Capital Medical University, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCRC-2021-01
Record Dates: First submitted 2022-01-25; First posted 2022-02-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Acute Ischemic Stroke; Mechanical Thrombectomy; Edaravone Dexborneol; Phase III
MeSH Terms: conditions — Ischemic Stroke | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Edaravone Dexborneol group (Experimental): Patients in this arm will be given Edaravone Dexborneol Concentrated Solution for injection twice a day for 10 to 14 days.
  Interventions: Drug: Edaravone Dexborneol Concentrated Solution for injection
- Edaravone Dexborneol Placebo group (Placebo Comparator): Patients in this arm will be given a placebo of Edaravone Dexborneol for injection twice a day for 10 to 14 days.
  Interventions: Drug: Edaravone Dexborneol placebo

INTERVENTIONS:
Drug: Edaravone Dexborneol Concentrated Solution for injection — Edaravone and Dexborneol Concentrated Solution for Injection, 15 ml (37.5 mg, containing edaravone 30 mg and dexborneol 7.5 mg) in 3 ampoule bottles, twice a day for 10 to 14 days.
  Other Names: Xian Bi Xin, CFDA Approval Number H20200007
  Arms: Edaravone Dexborneol group
Drug: Edaravone Dexborneol placebo — Edaravone and Dexborneol placebo, 15 ml in 3 ampoule bottles, twice a day for 10 to 14 days.
  Other Names: Xian Bi Xin placebo
  Arms: Edaravone Dexborneol Placebo group

SUMMARY:
This study is a multicentre, randomized, double-blind, placebo parallel controlled, investigator-sponsored study that aims to investigate the efficacy and safety of Edaravone Dexborneol treatment in patients with acute ischemic stroke who had received early reperfusion therapy.

DETAILED DESCRIPTION:
This is a multicentre, randomized, double-blind, placebo-controlled trial that aims to investigate the efficacy and safety of Edaravone Dexborneol treatment in patients with acute ischemic stroke who had received early reperfusion therapy. Patients who were eligible to the inclusion criteria and ineligible to the exclusion criteria will be randomly assigned into two groups by a 1:1 ratio after the ICF was received. Patients in one arm will be given 15 ml edaravone and dexborneol concentrated solution for injection (37.5 mg, containing edaravone 30 mg and dexborneol 7.5 mg) twice a day for 10-14 days, and those in the other arm will be given an equivalent placebo drug. All patients will be followed up for 90 days. The primary outcome is the proportion of modified Rankin Scale 0-2 and the safety outcome is the proportion of severe adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. 18 - 80 years, male or female;
2. Clinically diagnosed as acute anterior ischemic stroke, artery occlusion occurred at the terminal of the intracranial carotid artery, T-shaped bifurcation or M1 segment of the middle cerebral artery;
3. Within 24 hours of stroke onset;
4. Eligible for other imaging indications for bridging therapy or direct mechanical thrombectomy:

   ASPECTS ≥6 certified by the latest brain CT imaging; Patients within 6-16 hours after stroke onset should meet the mismatch criteria, which was defined as infarction core volume <70 ml, mismatch ratio ≥1.8 and the ischemic volume > 15 ml (DEFUSE-3 Criteria); or NIHSS score ≥ 10 with infarction -core volume < 31 cm3, or NIHSS score ≥ 20 with infarction core volume ≤ 51 cm3 (DAWN Criteria); Patients within 16-24 hours after stroke onset should meet the mismatch criteria, which was defined as NIHSS score ≥ 10 with infarction-core volume < 31 cm3, or NIHSS score ≥ 20 with infarction-core volume ≤ 51 cm3 (DAWN Criteria);
5. Planned to receive bridging therapy (endovascular therapy after intravenous alteplase) or direct endovascular therapy;
6. Pre-morbid modified Rankin Scale ≤1;
7. 6 ≤ NIHSS ≤ 25 before endovascular therapy;
8. Signed informed consent from subjects or legally authorized representatives

Exclusion Criteria:

1. CT indicates intracranial hemorrhagic diseases, such as hemorrhagic stroke, subdural hematoma, ventricular hemorrhage, or subarachnoid hemorrhage, etc.;
2. Had been given any intravenous thrombolytic drug other than alteplase before bridging therapy;
3. Hypersensitive to edaravone, (+)-2- dexborneol or auxiliary materials;
4. Prior receipt of edaravone or any other neuroprotective drugs;
5. History of congenital or acquired hemorrhagic disease, coagulation factor deficiency disease, or thrombocytopenic disease, etc.;
6. Systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥110 mmHg after antihypertensive treatment;
7. Serum alanine aminotransferase (ALT) or aspartate transaminase (AST) elevates over 3 times of upper limit of normal;
8. Recent or current serum creatinine is known to exceed 1.5 times the upper limit of normal, or estimated glomerular filtration rate (eGFR) < 60 mL/min;
9. Pregnancy, lactation, or planned pregnancy within 90 days;
10. Those who cannot complete informed consent or follow-up treatment due to severe mental disorder or dementia;
11. Those with a malignant tumor, severe systemic diseases, or predict survival time <90 days;
12. Participate in another interventional clinical study within 30 days before randomization or participate in another interventional clinical study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1362 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-05-19 (Actual)

PRIMARY OUTCOMES:
Favorable functional outcome | at 90 days after randomization
  Rate of favorable functional outcome defined as a modified Rankin Scale (mRS, scores range from 0 to 6, with 0 to 2 indicating favorable outcome and 3 to 6 indicating unfavorable outcome including 6 as death) score of 0-2
Incidence of severe adverse event (Safety outcome) | at 90 days after randomization
  The incidence of Severe Adverse Event (SAE) emerged during the whole study period

SECONDARY OUTCOMES:
Excellent functional outcome | at 90 days after randomization
  Rate of excellent functional outcome defined as a mRS score 0-1
NIHSS score change | at 10-14 days after randomization
  The change of NIHSS score defined as the NIHSS score of day 10-14 minus that of baseline
NIHSS score decreases ≥4 | at 10-14 days after randomization
  Defined as the proportion of patients with NIHSS score decrease ≥ 4 from day 10-14 to baseline
All-cause mortality | at 90 days after randomization
  All-cause mortality at 90 days after randomization
Symptomatic intracranial hemorrhage (sICH) | at 24-36 hours after randomization
  The proportion of patients who experienced sICH
Neurological deterioration | at day 1 after randomization
  Defined as the NIHSS score increases ≥4 from day 1 to baseline
Stroke recurrence | within 90 days after randomization
  Defined as a new ischemic or hemorrhagic stroke occurred within 90 days after randomization
Adverse events (AE) | within 90 days after randomization
  The proportion of patients who experienced AE

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, MD., Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hill MD, Goyal M, Menon BK, Nogueira RG, McTaggart RA, Demchuk AM, Poppe AY, Buck BH, Field TS, Dowlatshahi D, van Adel BA, Swartz RH, Shah RA, Sauvageau E, Zerna C, Ospel JM, Joshi M, Almekhlafi MA, Ryckborst KJ, Lowerison MW, Heard K, Garman D, Haussen D, Cutting SM, Coutts SB, Roy D, Rempel JL, Rohr AC, Iancu D, Sahlas DJ, Yu AYX, Devlin TG, Hanel RA, Puetz V, Silver FL, Campbell BCV, Chapot R, Teitelbaum J, Mandzia JL, Kleinig TJ, Turkel-Parrella D, Heck D, Kelly ME, Bharatha A, Bang OY, Jadhav A, Gupta R, Frei DF, Tarpley JW, McDougall CG, Holmin S, Rha JH, Puri AS, Camden MC, Thomalla G, Choe H, Phillips SJ, Schindler JL, Thornton J, Nagel S, Heo JH, Sohn SI, Psychogios MN, Budzik RF, Starkman S, Martin CO, Burns PA, Murphy S, Lopez GA, English J, Tymianski M; ESCAPE-NA1 Investigators. Efficacy and safety of nerinetide for the treatment of acute ischaemic stroke (ESCAPE-NA1): a multicentre, double-blind, randomised controlled trial. Lancet. 2020 Mar 14;395(10227):878-887. doi: 10.1016/S0140-6736(20)30258-0. Epub 2020 Feb 20. PMID 32087818
- [Background] Xu J, Wang A, Meng X, Yalkun G, Xu A, Gao Z, Chen H, Ji Y, Xu J, Geng D, Zhu R, Liu B, Dong A, Mu H, Lu Z, Li S, Zheng H, Chen X, Wang Y, Zhao X, Wang Y; TASTE Trial Investigatorsdagger. Edaravone Dexborneol Versus Edaravone Alone for the Treatment of Acute Ischemic Stroke: A Phase III, Randomized, Double-Blind, Comparative Trial. Stroke. 2021 Mar;52(3):772-780. doi: 10.1161/STROKEAHA.120.031197. Epub 2021 Feb 16. PMID 33588596
- [Derived] Wang C, Gu H, Huo X, Yuan B, Li S, Xu J, Jiang Y, Jing J, Yao X, Li Z, Long F, Ma Z, Zhuang X, Xu L, Jin Y, Huang W, Zhang Y, Wen J, Wang A, Pan Y, Ye W, Yu W, Cheng A, Wang M, Dong Q, Xu A, Wang N, Yang Y, Meng X, Liu L, Zhao X, Li H, Miao Z, Li Z, Wang Y; TASTE-2 investigators. Edaravone dexborneol versus placebo on functional outcomes in patients with acute ischaemic stroke undergoing endovascular thrombectomy (TASTE-2): randomised controlled trial. BMJ. 2026 Jan 7;392:e086850. doi: 10.1136/bmj-2025-086850. PMID 41500725